CLINICAL TRIAL: NCT04700826
Title: Preventing Stroke, Premature Death and Cognitive Decline in a Broader Community of Patients With Atrial Fibrillation Using Healthcare Data for Pragmatic Research: A Randomised Controlled Trial
Brief Title: Preventing Stroke, Premature Death and Cognitive Decline in a Broader Community of Patients With Atrial Fibrillation
Acronym: DaRe2THINK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Clinical Practice Research Datalink (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); University of Oxford (Other); London School of Economics and Political Science (Other); Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERN_20-1747; 290420 (Other: IRAS)
Record Dates: First submitted 2020-12-04; First posted 2021-01-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; anticoagulation; stroke; dementia
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Dementia | interventions — N(4)-oleylcytosine arabinoside; apixaban; Dabigatran; edoxaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Individual patient, open-label, event driven RCT with 1:1 allocation to DOAC or no additional therapy (usual care). Choice of DOAC (apixaban, dabigatran, edoxaban or rivaroxaban) according to local practice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Oral anticoagulants (DOAC) (Experimental): Commence DOAC even with low or intermediate risk of stroke or thromboembolism, which could include currently licensed drugs apixaban, dabigatran, edoxaban or rivaroxaban; choice of drug and dose according to local practice guidelines
  Interventions: Drug: Direct Oral Anticoagulants
- No anticoagulant therapy (usual care) (No Intervention): Continuation of usual anticoagulant prescribing practice in patients with AF; e.g. according to National Institute for Health and Care Excellence (NICE), patients with AF should commence oral anticoagulation with a CHA2DS2-VASc score of 2 or above.

INTERVENTIONS:
Drug: Direct Oral Anticoagulants — choice of DOAC (apixaban, dabigatran, edoxaban or rivaroxaban) according to local practice
  Other Names: apixaban, dabigatran, edoxaban or rivaroxaban
  Arms: Direct Oral anticoagulants (DOAC)

SUMMARY:
The DaRe2 approach (healthcare Data for pragmatic clinical Research in the NHS - primary 2 secondary) is designed to operationalise efficient, nationwide, primary care approaches for randomised trials embedded within the UK National Health Service (NHS), providing automated screening, targeted patient enrolment and 'no-visit' follow-up through innovations in big data and technology solutions.

DaRe2THINK will be the first exemplar of this system, and is appropriately focused on the intersection of key national priorities for healthcare; atrial fibrillation (a heart rhythm condition that will double in prevalence in the next few decades) and the impact this condition has on stroke, thromboembolic events, cognitive impairment and vascular dementia. The trial will test the hypothesis that direct oral anticoagulants (DOACs), now commonly used in older patients with atrial fibrillation (AF), are effective and cost-effective at reducing major adverse clinical events in younger patients at low or intermediate risk of stroke, and can reduce the high rate of cognitive decline. The health technology innovations noted above will allow the investigators to answer this important clinical question, as well as demonstrate the capacity and potential of this system for future, large-scale healthcare-embedded clinical trials for patient benefit.

DETAILED DESCRIPTION:
Designed with a Patient and Public Involvement Team, DaRe2THINK is an individual-patient, open-label, event-driven randomised trial with 1:1 allocation to DOAC or no additional therapy (usual care). Automated screening will occur of over 12 million patients in England, with targeted recruitment to practices with eligible patients, regular updates to General Practitioners, simple processes for centre inclusion and patient randomisation, remote e-consent and no additional visits for any patient. The primary outcome is a comprehensive composite of any thromboembolic event, ascertained entirely using electronic healthcare records within both primary and secondary NHS care across the nation. All endpoint data will follow a pre-published coding manual for extracted electronic healthcare data. The key secondary outcome is the change in patient-reported cognitive function, using remote technology solutions to save time for clinical staff and patients. DaRe2THINK will carefully assess and validate safety outcomes relating to major and minor bleeding. A systematic health economic analysis will determine NHS and societal cost-effectiveness of DOAC therapy in this younger population of patients with AF. DaRe2THINK will initially run over a 5-year period (outcomes as listed below), with longer-term outcomes (in particular cardiovascular death, cognitive function and vascular dementia) reassessed at 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AF (previous, current or chronic)
2. Age at enrolment ≥55 years to ≤73 years

Exclusion Criteria based on coding in Primary Care:

1. Prior documented stroke, transient ischaemic attack or systemic thromboembolism.
2. Combination of multiple known risk factors for stroke where oral anticoagulation would ordinarily be started, including: Heart failure; Hypertension; Age 65 years or older; Diabetes mellitus; Previous myocardial infarction, peripheral artery disease or aortic plaque; and/or Female gender.
3. Any prior history of intracranial bleeding.
4. Prior major bleeding requiring hospitalisation in the last 3 years.
5. Condition that poses a significant risk for bleeding (within 12 months) including gastrointestinal ulceration, brain/spinal/ophthalmic injury or surgery, arteriovenous malformations or vascular aneurysms, major intraspinal or intracerebral vascular abnormalities, hepatic disease associated with coagulopathy, known or suspected oesophageal varices, and cancers with high bleeding risk.
6. Estimated glomerular filtration rate <30 mL/min/1.73m2 measured within the last 12 months.
7. Patients receiving systemic treatment with azole-antimycotics within the last 3 months (ketoconazole, itraconazole, voriconazole and posaconazole).
8. Documented diagnosis of dementia.
9. Hypersensitivity or known intolerance to direct oral anticoagulants.

Exclusion criteria based on review by Primary Care staff:

1. Currently receiving an anticoagulant.
2. Any clinical indication for anticoagulation.
3. Active clinically-significant bleeding.
4. Life expectancy estimated <2 years.
5. Participant unable or unwilling to provide informed consent for access and linkage of past and future electronic healthcare records.
6. Currently participating in another clinical trial.
7. Women of childbearing potential.

Ages: 55 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint - Time to first event | 5 years
  Composite primary endpoint - Time to first event of cardiovascular mortality, ischaemic cerebrovascular events (stroke and transient ischaemic attacks), all thromboembolic events (including venous and arterial thromboembolism), myocardial infarction and vascular dementia

SECONDARY OUTCOMES:
Change in cognitive function using the UK Biobank fluid intelligence/reasoning test (mixed-effects repeated measures analysis) | 5 years
  Change in cognitive function using the UK Biobank fluid intelligence/reasoning test (mixed-effects repeated measures analysis)
Change in cognitive function using the UK Biobank trail making test (mixed-effects repeated measures analysis) | 5 years
  Change in cognitive function using the UK Biobank trail making test (mixed-effects repeated measures analysis)
Change in cognitive function using the UK Biobank symbol digit substitution test (mixed-effects repeated measures analysis) | 5 years
  Change in cognitive function using the UK Biobank symbol digit substitution test (mixed-effects repeated measures analysis)
. Change in cognitive function using the UK Biobank non-verbal fluid reasoning matrices test (mixed-effects repeated measures analysis) | 5 years
  . Change in cognitive function using the UK Biobank non-verbal fluid reasoning matrices test (mixed-effects repeated measures analysis)
Incremental cost per quality-adjusted life-years gained from the healthcare perspective. | 5 years
  Incremental cost per quality-adjusted life-years gained from the healthcare perspective.
Incremental cost per quality-adjusted life-years gained from the societal perspective. | 5 years
  Incremental cost per quality-adjusted life-years gained from the societal perspective.
Time to composite of major adverse cardiovascular events (non-fatal stroke, non-fatal myocardial infarction and cardiovascular death). | 5 years
  Time to composite of major adverse cardiovascular events (non-fatal stroke, non-fatal myocardial infarction and cardiovascular death).
Time to any major bleeding or clinically-relevant non-major bleeding that requires hospitalisation. | 5 years
  Time to any major bleeding or clinically-relevant non-major bleeding that requires hospitalisation.
Time to minor bleeding that requires attention from primary care (any bleeding that leads to a primary care consultation). | 5 years
  Time to minor bleeding that requires attention from primary care (any bleeding that leads to a primary care consultation).
Time to haemorrhagic stroke and other types of intracranial bleeding. | 5 years
  Time to haemorrhagic stroke and other types of intracranial bleeding.
Number of all-cause general practice visits. | 5 years
  Number of all-cause general practice visits.
Number of all-cause hospital admissions. | 5 years
  Number of all-cause hospital admissions.
Duration of all-cause hospital admissions. | 5 years
  Duration of all-cause hospital admissions.
Number of heart failure hospitalisations. | 5 years
  Number of heart failure hospitalisations.
Duration of heart failure hospitalisations. | 5 years
  Duration of heart failure hospitalisations.
Time to all-cause mortality. | 5 years
  Time to all-cause mortality.
Time to cardiovascular death | 5 years
  Time to cardiovascular death
Patient-reported quality of life using the Euroqol five-dimensions five-level (EQ-5D-5L) summary index score (mixed-effects repeated measures analysis) | 5 years
  Patient-reported quality of life using the Euroqol five-dimensions five-level (EQ-5D-5L) summary index score (mixed-effects repeated measures analysis) Range 0 = death to 1 = complete health
Patient-reported quality of life using the EQ-5D-5L visual analogue score (mixed-effects repeated measures analysis) | 5 years
  Patient-reported quality of life using the EQ-5D-5L visual analogue score (mixed-effects repeated measures analysis) Range 0-100, with a higer score indicating better quality of life.
Time to ischaemic cerebrovascular event (stroke and transient ischaemic attacks) | 5 years
  Time to ischaemic cerebrovascular event (stroke and transient ischaemic attacks)
Cumulative number of ischaemic cerebrovascular events (stroke and transient ischaemic attacks) | 5 years
  Cumulative number of ischaemic cerebrovascular events (stroke and transient ischaemic attacks)
Time to any thromboembolic event (including venous and arterial thromboembolism) | 5 years
  Time to any thromboembolic event (including venous and arterial thromboembolism)
Time to arterial thromboembolic event | 5 years
  Time to arterial thromboembolic event
Time to venous thromboembolic event | 5 years
  Time to venous thromboembolic event
Cumulative number of thromboembolic events (including venous and arterial thromboembolism) | 5 years
  Cumulative number of thromboembolic events (including venous and arterial thromboembolism)
Time to myocardial infarction | 5 years
  Time to myocardial infarction
Cumulative number of myocardial infarctions | 5 years
  Cumulative number of myocardial infarctions
Time to vascular dementia | 5 years
  Time to vascular dementia

OTHER OUTCOMES:
Potential participants located by CPRD | 5 years
  Number/proportion of potential participants located by CPRD and notified to the lead NIHR Clinical Research Network (CRN)
Primary care practices completing sign up | 5 years
  Number/proportion of primary care practices that have completed sign-up processes
Patients on automated screening successfully recruited | 5 years
  Number/proportion of patients eligible on automated screening that are successfully recruited
Rate of patient recruitment | 5 years
  Rate of patient recruitment
Patient reported compliance | 5 years
  Patient-reported compliance to DOAC therapy in the DOAC arm
Repeat prescriptions for DOAC | 5 years
  Repeat prescriptions obtained for DOAC therapy
Proportion of participant time-points with missing data for EQ-5D-5L patient-reported quality of life | 5 years
  Missing data rates for 6-monthly patient-reported Euroqol five-dimensions five-level (EQ-5D-5L) summary index score, with death equivalent to a score of zero
Proportion of participant time-points with missing data for cognitive function using the UK Biobank fluid intelligence/reasoning test | 5 years
  Missing data rates for yearly patient-reported cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Dipak Kotecha, Principal Investigator — University of Birmingham and University Hospitals Birmingham NHS Foundation Trust; John Camm, Study Chair — St George's University of London; Chair of DaRe2THINK Independent TSC; Marcus Flather, Study Chair — Norwich Medical School; Chaire of DaRe2THINK Independent DMC; David Shukla, Principal Investigator — Deputy CI; Lead for NIHR West Midlands Primary Care CRN Team
Locations (1):
- University Hospitals Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Mobley AR, Tica O, Okoth K, Ghosh RE, Myles P, Williams T, Haynes S, Nirantharakumar K, Shukla D, Kotecha D; DaRe2THINK Trial Committees. Systematic approach to outcome assessment from coded electronic healthcare records in the DaRe2THINK NHS-embedded randomized trial. Eur Heart J Digit Health. 2022 Sep 16;3(3):426-436. doi: 10.1093/ehjdh/ztac046. eCollection 2022 Sep. PMID 36712153
- [Background] Mobley AR, Subramanian A, Champsi A, Wang X, Myles P, McGreavy P, Bunting KV, Shukla D, Nirantharakumar K, Kotecha D. Thromboembolic events and vascular dementia in patients with atrial fibrillation and low apparent stroke risk. Nat Med. 2024 Aug;30(8):2288-2294. doi: 10.1038/s41591-024-03049-9. Epub 2024 Jun 5. PMID 38839900
- [Background] Champsi A, Mobley AR, Subramanian A, Nirantharakumar K, Wang X, Shukla D, Bunting KV, Molgaard I, Dwight J, Arroyo RC, Crijns HJGM, Guasti L, Lettino M, Lumbers RT, Maesen B, Rienstra M, Svennberg E, Tica O, Traykov V, Tzeis S, van Gelder I, Kotecha D. Gender and contemporary risk of adverse events in atrial fibrillation. Eur Heart J. 2024 Sep 29;45(36):3707-3717. doi: 10.1093/eurheartj/ehae539. PMID 39217497

DOCUMENTS (1):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT04700826/Prot_000.pdf